CLINICAL TRIAL: NCT01054352
Title: A Double-blind, Placebo-Controlled, Randomized, Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Food Effect, and Pharmacokinetics and Pharmacodynamics of JNJ-38224342 in Healthy Patients and in Healthy Patients With Seasonal Allergic Rhinitis
Brief Title: A Single and Multiple Dose Study to Explore the Safety of JNJ-38224342 in Healthy Patients and Patients With Seasonal Allergies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016798
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Seasonal allergies; Allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 001 (Experimental): JNJ38224342/placebo one of six (6) single ascending doses (25 100 300 600 1250 or 2000 mg) of JNJ 38224342 or matching placebo up to four (4) additional cohorts consisting of healthy male volunteers may be added
  Interventions: Drug: JNJ38224342/placebo
- 002 (Experimental): JNJ38224342/placebo multiple ascending oral doses (100 250 500 750 mg) of JNJ 38224342 or matching placebo administered for 14 consecutive days in healthy male or female volunteers.up to four (4) additional cohorts consisting of healthy male or female volunteers may be added
  Interventions: Drug: JNJ38224342/placebo
- 003 (Experimental): JNJ38224342 single oral 100mg dose of JNJ 38224342 as a solution versus a single oral dose of JNJ 38224342 as a capsule formulation with and without food in healthy male volunteers
  Interventions: Drug: JNJ38224342
- 004 (Experimental): JNJ38224342/placebo multiple oral doses of JNJ38224342 or matching placebo administered for up to 14 consecutive days in male and female volunteers number of days dosed and actual dose levels food requirements and regimens will be determined based on the data from Parts 1 2 and 3.
  Interventions: Drug: JNJ38224342/placebo

INTERVENTIONS:
Drug: JNJ38224342 — multiple ascending oral doses (100, 250, 500, 750 mg) of JNJ 38224342 or matching placebo, administered for 14 consecutive days in healthy male or female volunteers
  Arms: 003
Drug: JNJ38224342/placebo — up to four (4) additional cohorts consisting of healthy male volunteers may be added
  Arms: 002
Drug: JNJ38224342/placebo — .up to four (4) additional cohorts consisting of healthy male or female volunteers may be added
  Arms: 004
Drug: JNJ38224342/placebo — one of six (6) single ascending doses (25, 100, 300, 600, 1250 or 2000 mg) of JNJ 38224342 or matching placebo
  Arms: 001

SUMMARY:
A single and multiple dose study to assess the safety of JNJ 38224342 compared to placebo in healthy volunteers and in volunteers with seasonal allergies.

DETAILED DESCRIPTION:
A four-part, single and multiple dose study to investigate the safety of JNJ-38224342 versus placebo in healthy patients and in patients with seasonal allergies. Volunteers (or patients) are randomly assigned to one of four treatment groups or Parts. Part 1 and 2 are randomized (study drug will be assigned by chance) and double-blind (neither the physician nor volunteer knows the identity of the assigned drug). In Part 1 patients receive a single oral dose of either 25, 100, 300, 600, 1250 or 2000 mg of JNJ-38224342 or placebo. In Part 2 patients receive multiple oral doses of either 100, 250, 500 or 700 mg of JNJ-38224342 or placebo administered over 14 days. Part 3 (for male volunteers only) is open-label (all people involved know the identity of the assigned drug), 2-period crossover (meaning that volunteers will receive both treatments at different times) study of the effects of food on JNJ-38224342. Participants will be given a single 100 mg oral dose (either solution or capsule formulation). Part 4 is for patients with seasonal allergies only. The dose of JNJ-38224342 will be determined based on information collected in Parts 1 - 3. Patients that participate in part 4 of the study will also have their nasal passage flushed out with salt water and the contents will be collected. Patients will be asked to remain in the clinic for either 5 days or 18 days depending on what part of the study they are participating in. A physical exam will be performed and a medical history collected. Safety evaluations include adverse event monitoring, blood pressure measurements, ECG and lab work requiring blood and urine samples at various time points throughout the study. Single oral dose of either 25, 100, 300, 600, 1250 or 2000mg of JNJ-38224342 or placebo; Multiple oral dose of either 100, 250, 500 or 700 mg of JNJ-38224342 or placebo administered over 14 days; single oral 100mg dose of JNJ 38224342 as a solution versus capsule with or without food; multiple oral doses of JNJ38224342 or placebo administered for up to 14 days where the number of days dosed, actual dose levels, food requirements will be determined based on the data from Parts 1, 2, and 3

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers
* If male, willing to use an acceptable method of birth control for duration of study and for 90 days post study
* Females must be post menopausal, surgically sterilized and cannot be pregnant or lactating (all parts of study)
* Have a clinical history of allergic rhinitis during the ragweed pollen season and a positive skin test for ragweed allergy are required (for part 4 of study only)

Exclusion Criteria:

* Clinically significant medical illnesses, laboratory or ECG findings
* History of allergy to aspirin or nonsteroidal anti-inflammatory drugs
* history of alcohol or drug abuse within the last 5 years
* HIV or Hepatitis B or C positive
* Receipt of an investigational drug or use of an investigational medical device within the last month
* History of asthma or severe respiratory infection or disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 182 (Actual)
Dates: Start 2010-02; Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To assess safety and pharmacokinetics of single and multiple oral ascending doses of JNJ-38224342 with and without food in healthy volunteers and patients with seasonal allergies as determined by occurrence of adverse events, lab test results, vital sign | from the time of the first dose to 7-11 days after the last dose administered

SECONDARY OUTCOMES:
Evaluate the results of biomarker assessments performed during Parts 2 and 4 of the trial. | from 7-11 days post the last administered dose
Evaluate the effectiveness of treatment based on nasal symptoms for Part 4. | from 7-11 days post the last administered dose

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Mississauga, Ontario, Canada